CLINICAL TRIAL: NCT06740045
Title: Opening the "Black Box" on Tezepelumab's Effect on Chronic Rhinosinusitis With Severe Asthma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Andrew Thamboo, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Dr. Andrew Thamboo, MD, Clinical Assistant Professor, St. Paul's Sinus Centre
Organization: St. Paul's Sinus Centre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H24-02151
Record Dates: First submitted 2024-08-13; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Asthma; Chronic Rhinosinusitis With Nasal Polyps
MeSH Terms: conditions — Asthma | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: The proposed design is a 24-week pilot study to investigate the histo-inflammatory and remodeling profiles and clinical outcomes of Chronic Rhinosinusitis with Nasal Polyps (CRSwNP) patients with Severe Asthma (SA) treated with Tezepelumab. The investigators plan to recruit approximately 10 subjects with (CRSwNP) and severe asthma as a "proof of concept" study. Eligible subjects will be requested to participate in the study for a maximum of 24 weeks, during which subjects will remain on their existing standard of care therapy. At Visit 2 (week 0), subjects will receive either add-on Tezepelumab (210 mg) during the 24-week treatment period. Study medication will be administered subcutaneously (SC) every 4 weeks for a total of 6 doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tezepelumab (Experimental): Tezepelumab 210 mg subcutaneous injection every 4 weeks to all 10 participants
  Interventions: Biological: Tezepelumab

INTERVENTIONS:
Biological: Tezepelumab — 10 patients will receive teszpire
  Other Names: Teszpire

SUMMARY:
The study explores how chronic rhinosinusitis (CRS) and asthma share a common inflammatory process, particularly affecting patients with both conditions. Interaction between immune cells (Interleukins) and Th2 cytokines, such as TSLP, exacerbates asthma control in CRS patients, especially those with nasal polyps (CRSwNP). TSLP plays a pivotal role in initiating and maintaining airway inflammation in both diseases. Tezepelumab, a biologic therapy targeting TSLP, shows promise in reducing inflammation markers in severe asthma but its impact on CRSwNP and quality of life remains unclear. The study proposes investigating Tezepelumab's efficacy in treating CRSwNP and severe asthma to inform future biologic therapies.

DETAILED DESCRIPTION:
The investigators hypothesize that TSLP blockade with Tezepelumab will a) reduce upper airway inflammation based on histological, inflammatory, and remodeling biomarkers, that are evident in the airway remodeling process and b) correlate to a positive clinical response. Thus, nasal samples from chronic rhinosinusitis with nasal polyps (CRSwNP) patients with Severe Asthma (SA) pre- and post-treatment will exhibit inflammatory biomarkers and histopathological evidence that could prove responsive to the Tezepelumab.

The overall research objectives are to evaluate the effect of study intervention (Tezepelumab) on CRSwNP-SA outcomes through a) evaluating the sinonasal inflammatory profile, histopathological features, and remodeling biomarkers and b) investigating the impact of Tezepelumab on the CRSwNP-related clinical outcomes in the treated study subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must be ≥19 of age at the time of signing the informed consent form
* Capable of giving signed informed consent.
* Having CRSwNP based on clinical symptoms and/or radiographic or endoscopic evidence of inflammation in their upper airways (Diagnosis consistent with EPOS 2020)(2)and severe asthma:

  * SA based on GINA criteria (37) and confirmed with spirometry and assessmenton the previous history of asthma (a pre-post bronchodilator spirometry ormethacholine challenge to document the positive or negative history of asthmawill be performed if there is no clinical record).
  * Nasal polyp score (NPS) of at least 2 on each side
* Females of childbearing potential must commit using an acceptable method of birthcontrol for the duration of the study and they must have a negative urine pregnancy test ateach study visit
* Not expecting to have surgery within the next 7 months

Exclusion Criteria:

* Have previously undergone sinus surgery or nasal polypectomy
* A history of organ transplantation such as lung transplantation
* Previously or currently using immunomodulator medications or antihistamines
* A history of auto-immune diseases
* Current or past sinonasal or bronchial tumors
* Currently using systemic or oral corticosteroids
* Women who are pregnant, plan to become pregnant, or breastfeed during the trial
* Current participation in any other interventional treatment trials
* Compliance: is unlikely to comply with study visits based on investigator judgment:
* Diagnosed or suspected malignant or premalignant nasal disease (e.g. SchniderianPapilloma, unilateral nasal polyposis)
* Fungal rhinosinusitis (CT/Histology), positive Aspergillus skin prick testing and/orpositive Aspergillus IgE RAST (Radioallergosorbent) testing
* Malignant neoplasm within 5 years (from screening) excluding basal cell or squamouscell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterinecervix treated locally and without metastatic disease for 3 years.
* Active bleeding disorders, and/or inability to support interruption to anticoagulant or anti-platelet therapies for nasal biopsy.
* Severe nasal deformity precluding endoscopic assessment/biopsy of postnasal space
* Have an acute or chronic infection (excluding that related to CRS) requiring managementas follows:

  * Currently on any treatment for a chronic infection such as pneumocystis,cytomegalovirus, herpes simplex virus, herpes zoster, or atypical mycobacteria
  * Hospitalisation solely for the treatment of proven infection requiring parenteral (IV orIM) antibiotics (antibacterial, antiviral, antifungal, or anti-parasitic agents) within 60days of Day 1
  * Proven severe infection requiring outpatient treatment with parenteral (IV or IM)antibiotics (antibacterial, antiviral, antifungal, or anti-parasitic agents) within 60 daysof Day 1. Prophylactic anti-infective treatment is allowed.
* Known positive human immunodeficiency virus (HIV) status
* Known positive Hepatitis B (HB) or Hepatitis C status
* Have clinical evidence of significant unstable or uncontrolled acute or chronic diseaseswhich, in the opinion of the principal investigator, could confound the results of the study orput the participant at undue risk
* Have a planned surgical procedure, laboratory abnormality, or condition that, in theopinion of the principal investigator, makes the participant unsuitable for the study.
* Have received any investigational agent (that is not approved for sale in Canada) within60 days of Day 1
* Smoking history; current or former smokers with a smoke history of packs year >15
* Subjects with parasitic (helminthic) infection
* Subjects with hypersensitivity; with allergy/intolerance to a monoclonal antibody or biologics
* Subjects allergic to Aspirin (ASA) and non-steroidal anti-inflammatory drugs (NSAIDs)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Eosinophil Count | From baseline to 24 weeks
  Measurement of eosinophil count in tissue samples. Cells per high power field (HPF) or cells per millimeter squared (cells/mm²).
Neutrophil count | From baseline to 24 weeks.
  Measurement of neutrophil count in tissue samples. Cells per high power field (HPF) or cells per millimeter squared (cells/mm²).
Basement Membrane Thickness | From baseline to 24 weeks
  Measurement of the thickness of the basement membrane in tissue samples. Micrometers (µm)
Fibrosis | From baseline to 24 weeks
  Assessment of the extent of fibrosis in tissue samples, which may involve scoring systems or quantitative measurements
Squamous Metaplasia | From baseline to 24 weeks
  Immunohistochemical staining will be used to identify the presence of squamous metaplasia, with scoring based on percentage of positive cells.
Lymphocytic Proliferation | From baseline to 24 weeks
  Lymphocytic proliferation will be assessed using immunohistochemistry (IHC) to measure the Ki-67 proliferation index in tissue samples, specifically identifying the percentage of Ki-67-positive lymphocytes

SECONDARY OUTCOMES:
Immunoglobulin leves | 24 weeks
  IgE, IgG, IgA,
Th2 Cytokines | 24 weeks
  Measurement of Th2 cytokines such as IL-4, IL-5, IL-13
Th1/Th17 Cytokines | 24 weeks
  Measurement of Th1/Th17 cytokines such as IFN-γ and IL-17.
Myeloperoxidase (MPO) | 24 weeks
  Measurement of MPO levels in sinonasal samples or serum.
Interferon-γ (IFN-γ) | 24 weeks
  Measurement of IFN-γ levels in sinonasal samples or serum.
SNOT-22 (Sino-Nasal Outcome Test 22-item) | 24 weeks
  Assessment of sinonasal symptoms and their impact on quality of life using a 22-item questionnaire.
Health-Related Quality of Life | 24 weeks
  Measurement of health-related quality of life using the EuroQualityOfLife 5-Dimension 5-Level (EQ-5D-5L) instrument.
  The EQ-5D-5L includes 5 dimensions of health (Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression) with 5 levels of severity for each dimension (no problems, slight problems, moderate problems, severe problems, and extreme problems).
  For the overall EQ-5D-5L index score, it typically ranges from:
  Minimum Value: 0 (representing death) Maximum Value: 1 (representing perfect health) In some versions, a negative score can be obtained, which represents a state "worse than death."
Asthma Control Questionnaire | 24 weeks
  Asthma control will be assessed using the 5-question Asthma Control Questionnaire (ACQ-5), which includes the following domains: symptoms, reliever medication use, and limitations on daily activities. Each question is rated on a scale from 0 (no symptoms) to 6 (maximum symptoms). The total score is the sum of the individual responses, with possible scores ranging from 0 to 30
Epithelial Changes | 24 weeks
  Measurement of epithelial changes in sinonasal tissues, including alterations in epithelial thickness, cell type, and structural modifications.
Modified Lund-Kennedy Endoscopy Score | 24 weeks
  Evaluation of sinonasal pathology using the Modified Lund-Kennedy endoscopy scoring system, which assesses factors like nasal polyp size, discharge, and mucosal appearance. Typically ranges from 0 to 24, where higher scores indicate more severe disease.
Lund-Mackay CT Scan Score | 24 weeks
  Evaluation of sinus opacifications and other CT scan findings using the Lund-Mackay scoring system, which assesses the extent of sinus disease. Typically ranges from 0 to 24. 0 (no opacification) to 2 (complete opacification)
Changes in smell | 24 weeks
  Measurement of changes in olfactory function using the University of Pennsylvania Smell Identification Test (UPSIT)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Thamboo, Principal Investigator — St Paul's Sonis Centre Director

IPD SHARING:
Plan to Share IPD: No